CLINICAL TRIAL: NCT03075306
Title: Randomized Trial of a Healthy Weight Intervention for Youth With Serious Emotional Disturbance
Acronym: CHAMPION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00130511; MH110968 (Other: National Institute of Mental Health)
Record Dates: First submitted 2017-03-04; First posted 2017-03-09 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss | interventions — Methods

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- usual care (No Intervention): usual care and materials on healthy weight
- intervention (Experimental): the 12-month CHAMPION intervention with a health coach who provides healthy lifestyle counseling and support for weight management, a healthy diet and increased physical activity incorporating techniques to engage both the youth and parents
  Interventions: Behavioral: intervention

INTERVENTIONS:
Behavioral: intervention — the 12-month CHAMPION intervention with a health coach who provides healthy lifestyle counseling and support for weight management, a healthy diet and increased physical activity incorporating techniques to engage both the youth and parents
  Arms: intervention

SUMMARY:
The prevalence of overweight and obesity in youth with serious emotional disturbance (SED) exceeds the epidemic levels of overweight and obesity for children in the general population. Associated cardiovascular (CVD) risk factors such as glucose intolerance, hypertension and lipid abnormalities frequently already exist in obese children. Thus, focusing on overweight/obesity in youth with SED is critical to prevent their premature CVD. In 2015 the American Heart Association called attention to mental illnesses in youth as important risk conditions for early CVD and declared the need for transformational change in screening and management of overweight and obesity. Despite this, studies of healthy weight interventions in youth with SED are noticeably absent, and interventions will likely need to be tailored for this population who frequently have impulsivity, oppositional behavior and/or mood symptoms. In the general population, successful interventions targeting youth obesity often include active parental participation. Community mental health programs serving youth typically engage parents as part of routine treatment and therefore provide an unappreciated but potentially important opportunity to address overweight and obesity. The objective of this study is to design and rigorously test an innovative, scalable healthy weight intervention in youth with SED that incorporates parental engagement and provider support. The CHAMPION Trial is a two-arm trial partnering with community mental health organizations in Maryland. We will perform population-based screening to identify youth with overweight and obesity, and recruit and enroll 120 ages 8-18 years with SED with a BMI at or above the 85th%tile. The study will stratify by sex and site and randomly assign participants to receive a) usual care plus educational materials on healthy weight, or b) the 12-month CHAMPION intervention with a health coach who provides healthy lifestyle counseling and support for weight management, a healthy diet and increased physical activity incorporating techniques to engage both the youth and parents. The intervention's first 6 months will include frequent contacts, followed by a 6-month maintenance phase. The primary outcome will be decreased BMI z-score compared to control at 12 months; secondary outcomes include waist circumference, blood pressure, glucose, lipid levels, quality of life, and psychiatric symptoms at 6 and 12 mo. Antecedents of CVD begin early in youth, and those with SED are at particularly high risk. Breaking this cascade of risk factors leading to premature CVD will require capitalizing on the window of opportunity to intervene on overweight and obesity in youth with SED. The CHAMPION Trial will test an innovative, yet practical approach that could be readily incorporated into overall care of youth with SED.

ELIGIBILITY:
Inclusion Criteria:

* Ages 8 through 18 years

  * Measured BMI ≥ 85th percentile for age and sex
  * Currently receiving specialty mental health outpatient treatment
  * Consent by parent and assent by child
  * Completion of baseline data collection
  * Willing to accept randomization, and to participate in the intervention

Exclusion Criteria:

* Does not speak or understand English
* Developmental delay precluding integrity or completion of study procedures
* Primary 1 °substance-related disorders unless co-occur with another DSM mental or emotional disorder
* Serious health condition or medical disability likely to hinder accurate measurement of weight, for which weight loss is contraindicated (e.g. bulimia nervosa) or which would likely cause weight loss
* Prader-Willi Syndrome or other similar genetic disorder of obesity
* Weight greater than 400 pounds
* Chronic or repetitive use of non-psychiatric medications likely to cause weight gain or prevent weight loss (e.g., corticosteroids)
* Weight loss (>=5% of body weight) within last 6 months
* Pregnant or nursing.
* Planning to leave clinic within 6 mo. or move out of area within 12 mo.
* Investigator discretion

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 112 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2021-02-19 (Actual); Study Completion 2021-02-19 (Actual)

PRIMARY OUTCOMES:
BMI Z score | 12 months
  body mass index Z score

CONTACTS AND LOCATIONS:
Overall Officials: Gaul Daumit, MD, MHS, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Children's Mental Health Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
via NIMH